CLINICAL TRIAL: NCT00891696
Title: Nutritional and Contractile Regulation of Muscle Growth (Cycle 2)
Brief Title: Nutritional and Contractile Regulation of Muscle Growth
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Basic Science
Other Study IDs: 08-306; R01AR049877 (NIH)
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2015-06

CONDITIONS: Sarcopenia
Keywords: Sarcopenia; Aging; Metabolism; Muscle; mTOR; Essential Amino Acids; Exercise; Rapamycin
MeSH Terms: conditions — Sarcopenia; Motor Activity | interventions — Sirolimus; Nitroprusside

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (14):
- Exp 1: AA + Rap (Active Comparator): Participants will receive amino acid supplementation and rapamycin.
  Interventions: Drug: Rapamycin; Other: Amino acid supplementation
- Exp 1: AA (Placebo Comparator): Participants will receive amino acid supplementation and placebo rapamycin.
  Interventions: Other: Amino acid supplementation
- Exp 1: HEx + Rap (Active Comparator): Participants will receive rapamycin and placebo amino acid supplementation, and they will undergo high-intensity resistance exercise.
  Interventions: Drug: Rapamycin; Other: Low-intensity resistance exercise
- Exp 1: HEx (Placebo Comparator): Participants will receive placebo amino acid supplementation and placebo rapamycin, and they will undergo high-intensity resistance exercise.
  Interventions: Other: Low-intensity resistance exercise
- Exp 1: HEx + AA + Rap (Active Comparator): Participants will receive amino acid supplementation and rapamycin, and they will undergo high-intensity resistance exercise.
  Interventions: Drug: Rapamycin; Other: Amino acid supplementation; Other: Low-intensity resistance exercise
- Exp 1: HEx + AA (Placebo Comparator): Participants will receive amino acid supplementation and placebo rapamycin, and they will undergo high-intensity resistance exercise.
  Interventions: Other: Amino acid supplementation; Other: Low-intensity resistance exercise
- Exp 2: LExFR + Rap (Active Comparator): Participants will receive rapamycin and will undergo low-intensity resistance exercise with blood flow restriction.
  Interventions: Drug: Rapamycin; Device: Blood flow restriction cuff; Other: Low-intensity resistance exercise
- Exp 2 and 3: LExFR (Placebo Comparator): Participants will receive placebo rapamycin and will undergo low-intensity resistance exercise with blood flow restriction.
  Interventions: Device: Blood flow restriction cuff; Other: Low-intensity resistance exercise
- Exp 2: SNP (Active Comparator): Participants will receive sodium nitroprusside in a resting state.
  Interventions: Drug: Sodium nitroprusside
- Exp 2: FR (Active Comparator): Participants will undergo blood flow restriction in a resting state.
  Interventions: Device: Blood flow restriction cuff
- Exp 2: LEx + SNP (Active Comparator): Participants will receive sodium nitroprusside and undergo low-intensity resistance exercise.
  Interventions: Drug: Sodium nitroprusside; Other: Low-intensity resistance exercise
- Exp 3: LEx (Placebo Comparator): Participants will undergo low-intensity resistance exercise.
  Interventions: Other: Low-intensity resistance exercise
- Exp 3: HEx (Active Comparator): Participants will undergo high-intensity resistance exercise.
  Interventions: Other: Low-intensity resistance exercise
- Exp 3: HEx + AA (Active Comparator): Participants will receive amino acid supplementation and will undergo high-intensity resistance exercise.
  Interventions: Other: Low-intensity resistance exercise

INTERVENTIONS:
Drug: Rapamycin — Single 16-mg oral dose
  Arms: Exp 1: AA + Rap; Exp 1: HEx + AA + Rap; Exp 1: HEx + Rap; Exp 2: LExFR + Rap
Other: Amino acid supplementation — Nutritional drink containing essential amino acids
  Arms: Exp 1: AA; Exp 1: AA + Rap; Exp 1: HEx + AA; Exp 1: HEx + AA + Rap
Other: Low-intensity resistance exercise — Leg extension exercises on a Cybex leg extension machine
  Arms: Exp 1: HEx; Exp 1: HEx + AA; Exp 1: HEx + AA + Rap; Exp 1: HEx + Rap; Exp 3: HEx; Exp 3: HEx + AA
Drug: Sodium nitroprusside — Variable rate for 3 hours
  Arms: Exp 2: LEx + SNP; Exp 2: SNP
Device: Blood flow restriction cuff — Blood flow restriction for 5 minutes after the second biopsy
  Other Names: KAATSU cuff
  Arms: Exp 2 and 3: LExFR; Exp 2: FR; Exp 2: LExFR + Rap
Other: Low-intensity resistance exercise — Leg extension exercises on a Cybex leg extension machine
  Arms: Exp 2 and 3: LExFR; Exp 2: LEx + SNP; Exp 2: LExFR + Rap; Exp 3: LEx

SUMMARY:
Muscle wasting, which involves the loss of muscle tissue, is common in many conditions, such as cancer, AIDS, trauma, kidney failure, bone fracture, and sepsis. It is also prevalent among the elderly and in people who experience periods of physical inactivity and weightlessness. Muscle wasting can lead to overall weakness, immobility, physical dependence, and a greater risk of death when exposed to infection, surgery, or trauma. There is a need to develop scientifically based treatments that prevent muscle wasting. As one step towards such a goal, this study will examine the physiological and cellular mechanisms that regulate skeletal muscle growth.

DETAILED DESCRIPTION:
Skeletal muscle comprises about 40% of one's body weight and contains about 50% to 75% of all the proteins in the human body. The turnover of protein is a regular process in the human body. In healthy adults, the interplay between muscle protein synthesis and muscle protein breakdown results in no net growth or loss of muscle mass. But when the scale tips towards muscle protein breakdown, muscle wasting can occur. This can result in negative consequences, because not only does muscle fill the obvious role of converting chemical energy into mechanical energy for moving and maintaining posture, but muscle is also involved in the following less apparent roles: regulating metabolism; removing potentially toxic substances from blood circulation; producing fuel for other tissues; storing energy and nitrogen, both of which are important for fueling the brain and immune system; and facilitating wound healing during malnutrition, starvation, injury, and disease. Therefore, muscle is important not only for physical independence but also for mere survival of the human body. In fact, a mere 30% loss of the body's proteins results in impaired respiration and circulation and can eventually lead to death. The purpose of this study is to examine the physiological and cellular mechanisms that regulate skeletal muscle growth. Results from the study may help to develop future treatments for maintaining and possibly increasing muscle mass as a way to improve function, reduce disease complications, and increase survival.

This study will enroll healthy participants who will be randomly assigned to one of several treatment arms within one of three separate experiments. Overall, the three experiments will examine the following: (1) whether the mammalian target of rapamycin (mTOR) signaling pathway--a group of molecules that work together to control a specific cellular function--is responsible for stimulating muscle protein synthesis after resistance exercise and/or ingestion of an amino acid supplement; (2) whether restricting blood flow with a blood pressure cuff during low-intensity resistance exercise ultimately leads to muscle protein synthesis; and (3) whether aging is associated with reduced physiological and cellular mechanisms that are related to muscle protein synthesis and whether such a reduction can be overcome by post-exercise ingestion of an amino acid supplement or blood flow restriction during low-intensity resistance exercise.

Depending on which treatment arm participants are assigned to, they may receive amino acid supplementation, the drug rapamycin, the drug sodium nitroprusside, and/or placebo. They may also undergo high-intensity resistance exercise, low-intensity resistance exercise, or low-intensity resistance exercise along with blood flow restriction. All participants will attend a single 8-hour study visit and a follow-up visit 1 week later. During the study visit, participants will undergo the following: measurements of vital signs, height, and weight; blood and urine sampling; a dual energy x-ray absorptiometry (DEXA) scan; and an infusion study that will include additional blood sampling, muscle biopsies, and assigned interventions. The follow-up visit will include evaluation of any incisions that were made during the infusion study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 35 years of age for the young groups
* 60 to 85 years of age for the older groups
* In the follicular phase for the young women participants
* Ability to sign consent form, as based on a score of greater than 25 on the 30-item Mini Mental State Examination (MMSE)
* Stable body weight for at least 1 year

Exclusion Criteria:

* Physical dependence or frailty, as determined by impairment in any of the activities of daily living (ADLs), history of more than two falls per year, or significant weight loss in the past year
* Exercise training that consists of more than two weekly sessions of moderate to high intensity aerobic or resistance exercise
* Significant heart, liver, kidney, blood, or respiratory disease
* Peripheral vascular disease
* Diabetes mellitus or other untreated endocrine disease
* Active cancer
* History of cancer for participants who may be randomly assigned to rapamycin)
* Acute infectious disease or history of chronic infections (e.g., tuberculosis, hepatitis, HIV, herpes)
* Treatment with anabolic steroids or corticosteroids within 6 months of study entry
* Alcohol or drug abuse
* Tobacco use (smoking or chewing)
* Malnutrition (e.g., body mass index [BMI] less than 20 kg/m2, hypoalbuminemia, and/or hypotransferrinemia)
* Obesity (BMI greater than 30 kg/m2)
* Lower than normal hemoglobin levels

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2009-04; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis | Measured during the 8-hour infusion study

SECONDARY OUTCOMES:
Phosphorylation status of mTOR signaling proteins | Measured during the 8-hour infusion study

CONTACTS AND LOCATIONS:
Overall Officials: Blake Rasmussen, PhD, Principal Investigator — The University of Texas Medical Branch, Galveston
Locations (1):
- Department of Nutrition & Metabolism, University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fujita S, Dreyer HC, Drummond MJ, Glynn EL, Volpi E, Rasmussen BB. Essential amino acid and carbohydrate ingestion before resistance exercise does not enhance postexercise muscle protein synthesis. J Appl Physiol (1985). 2009 May;106(5):1730-9. doi: 10.1152/japplphysiol.90395.2008. Epub 2008 Jun 5. PMID 18535123
- [Result] Volpi E, Chinkes DL, Rasmussen BB. Sequential muscle biopsies during a 6-h tracer infusion do not affect human mixed muscle protein synthesis and muscle phenylalanine kinetics. Am J Physiol Endocrinol Metab. 2008 Oct;295(4):E959-63. doi: 10.1152/ajpendo.00671.2007. Epub 2008 Aug 19. PMID 18713956
- [Result] Drummond MJ, Miyazaki M, Dreyer HC, Pennings B, Dhanani S, Volpi E, Esser KA, Rasmussen BB. Expression of growth-related genes in young and older human skeletal muscle following an acute stimulation of protein synthesis. J Appl Physiol (1985). 2009 Apr;106(4):1403-11. doi: 10.1152/japplphysiol.90842.2008. Epub 2008 Sep 11. PMID 18787087
- [Result] Drummond MJ, McCarthy JJ, Fry CS, Esser KA, Rasmussen BB. Aging differentially affects human skeletal muscle microRNA expression at rest and after an anabolic stimulus of resistance exercise and essential amino acids. Am J Physiol Endocrinol Metab. 2008 Dec;295(6):E1333-40. doi: 10.1152/ajpendo.90562.2008. Epub 2008 Sep 30. PMID 18827171
- [Result] Drummond MJ, Fry CS, Glynn EL, Dreyer HC, Dhanani S, Timmerman KL, Volpi E, Rasmussen BB. Rapamycin administration in humans blocks the contraction-induced increase in skeletal muscle protein synthesis. J Physiol. 2009 Apr 1;587(Pt 7):1535-46. doi: 10.1113/jphysiol.2008.163816. Epub 2009 Feb 2. PMID 19188252
- [Result] Drummond MJ, Glynn EL, Fry CS, Dhanani S, Volpi E, Rasmussen BB. Essential amino acids increase microRNA-499, -208b, and -23a and downregulate myostatin and myocyte enhancer factor 2C mRNA expression in human skeletal muscle. J Nutr. 2009 Dec;139(12):2279-84. doi: 10.3945/jn.109.112797. Epub 2009 Oct 14. PMID 19828686
- [Result] Dreyer HC, Fujita S, Glynn EL, Drummond MJ, Volpi E, Rasmussen BB. Resistance exercise increases leg muscle protein synthesis and mTOR signalling independent of sex. Acta Physiol (Oxf). 2010 May;199(1):71-81. doi: 10.1111/j.1748-1716.2010.02074.x. Epub 2010 Jan 12. PMID 20070283
- [Result] Fry CS, Glynn EL, Drummond MJ, Timmerman KL, Fujita S, Abe T, Dhanani S, Volpi E, Rasmussen BB. Blood flow restriction exercise stimulates mTORC1 signaling and muscle protein synthesis in older men. J Appl Physiol (1985). 2010 May;108(5):1199-209. doi: 10.1152/japplphysiol.01266.2009. Epub 2010 Feb 11. PMID 20150565
- [Result] Drummond MJ, Glynn EL, Fry CS, Timmerman KL, Volpi E, Rasmussen BB. An increase in essential amino acid availability upregulates amino acid transporter expression in human skeletal muscle. Am J Physiol Endocrinol Metab. 2010 May;298(5):E1011-8. doi: 10.1152/ajpendo.00690.2009. Epub 2010 Feb 9. PMID 20304764
- [Result] Glynn EL, Fry CS, Drummond MJ, Dreyer HC, Dhanani S, Volpi E, Rasmussen BB. Muscle protein breakdown has a minor role in the protein anabolic response to essential amino acid and carbohydrate intake following resistance exercise. Am J Physiol Regul Integr Comp Physiol. 2010 Aug;299(2):R533-40. doi: 10.1152/ajpregu.00077.2010. Epub 2010 Jun 2. PMID 20519362
- [Result] Glynn EL, Fry CS, Drummond MJ, Timmerman KL, Dhanani S, Volpi E, Rasmussen BB. Excess leucine intake enhances muscle anabolic signaling but not net protein anabolism in young men and women. J Nutr. 2010 Nov;140(11):1970-6. doi: 10.3945/jn.110.127647. Epub 2010 Sep 15. PMID 20844186
- [Result] Drummond MJ, McCarthy JJ, Sinha M, Spratt HM, Volpi E, Esser KA, Rasmussen BB. Aging and microRNA expression in human skeletal muscle: a microarray and bioinformatics analysis. Physiol Genomics. 2011 May 1;43(10):595-603. doi: 10.1152/physiolgenomics.00148.2010. Epub 2010 Sep 28. PMID 20876843
- [Result] Dickinson JM, Fry CS, Drummond MJ, Gundermann DM, Walker DK, Glynn EL, Timmerman KL, Dhanani S, Volpi E, Rasmussen BB. Mammalian target of rapamycin complex 1 activation is required for the stimulation of human skeletal muscle protein synthesis by essential amino acids. J Nutr. 2011 May;141(5):856-62. doi: 10.3945/jn.111.139485. Epub 2011 Mar 23. PMID 21430254
- [Result] Drummond MJ, Fry CS, Glynn EL, Timmerman KL, Dickinson JM, Walker DK, Gundermann DM, Volpi E, Rasmussen BB. Skeletal muscle amino acid transporter expression is increased in young and older adults following resistance exercise. J Appl Physiol (1985). 2011 Jul;111(1):135-42. doi: 10.1152/japplphysiol.01408.2010. Epub 2011 Apr 28. PMID 21527663
- [Result] Fry CS, Drummond MJ, Glynn EL, Dickinson JM, Gundermann DM, Timmerman KL, Walker DK, Dhanani S, Volpi E, Rasmussen BB. Aging impairs contraction-induced human skeletal muscle mTORC1 signaling and protein synthesis. Skelet Muscle. 2011 Mar 2;1(1):11. doi: 10.1186/2044-5040-1-11. PMID 21798089
- [Result] Gundermann DM, Fry CS, Dickinson JM, Walker DK, Timmerman KL, Drummond MJ, Volpi E, Rasmussen BB. Reactive hyperemia is not responsible for stimulating muscle protein synthesis following blood flow restriction exercise. J Appl Physiol (1985). 2012 May;112(9):1520-8. doi: 10.1152/japplphysiol.01267.2011. Epub 2012 Feb 23. PMID 22362401
- [Result] Walker DK, Fry CS, Drummond MJ, Dickinson JM, Timmerman KL, Gundermann DM, Jennings K, Volpi E, Rasmussen BB. PAX7+ satellite cells in young and older adults following resistance exercise. Muscle Nerve. 2012 Jul;46(1):51-9. doi: 10.1002/mus.23266. Epub 2012 May 29. PMID 22644638
- [Result] Dickinson JM, Drummond MJ, Coben JR, Volpi E, Rasmussen BB. Aging differentially affects human skeletal muscle amino acid transporter expression when essential amino acids are ingested after exercise. Clin Nutr. 2013 Apr;32(2):273-80. doi: 10.1016/j.clnu.2012.07.009. Epub 2012 Aug 1. PMID 22889597
- [Result] Fry CS, Drummond MJ, Lujan HL, DiCarlo SE, Rasmussen BB. Paraplegia increases skeletal muscle autophagy. Muscle Nerve. 2012 Nov;46(5):793-8. doi: 10.1002/mus.23423. PMID 23055316
- [Result] Fry CS, Drummond MJ, Glynn EL, Dickinson JM, Gundermann DM, Timmerman KL, Walker DK, Volpi E, Rasmussen BB. Skeletal muscle autophagy and protein breakdown following resistance exercise are similar in younger and older adults. J Gerontol A Biol Sci Med Sci. 2013 May;68(5):599-607. doi: 10.1093/gerona/gls209. Epub 2012 Oct 22. PMID 23089333
- [Result] Reidy PT, Walker DK, Dickinson JM, Gundermann DM, Drummond MJ, Timmerman KL, Fry CS, Borack MS, Cope MB, Mukherjea R, Jennings K, Volpi E, Rasmussen BB. Protein blend ingestion following resistance exercise promotes human muscle protein synthesis. J Nutr. 2013 Apr;143(4):410-6. doi: 10.3945/jn.112.168021. Epub 2013 Jan 23. PMID 23343671
- [Result] Glynn EL, Fry CS, Timmerman KL, Drummond MJ, Volpi E, Rasmussen BB. Addition of carbohydrate or alanine to an essential amino acid mixture does not enhance human skeletal muscle protein anabolism. J Nutr. 2013 Mar;143(3):307-14. doi: 10.3945/jn.112.168203. Epub 2013 Jan 23. PMID 23343676
- [Result] Drummond MJ, Dickinson JM, Fry CS, Walker DK, Gundermann DM, Reidy PT, Timmerman KL, Markofski MM, Paddon-Jones D, Rasmussen BB, Volpi E. Bed rest impairs skeletal muscle amino acid transporter expression, mTORC1 signaling, and protein synthesis in response to essential amino acids in older adults. Am J Physiol Endocrinol Metab. 2012 May 15;302(9):E1113-22. doi: 10.1152/ajpendo.00603.2011. Epub 2012 Feb 14. PMID 22338078
- [Result] Paddon-Jones D, Rasmussen BB. Dietary protein recommendations and the prevention of sarcopenia. Curr Opin Clin Nutr Metab Care. 2009 Jan;12(1):86-90. doi: 10.1097/MCO.0b013e32831cef8b. PMID 19057193
- [Result] Drummond MJ, Dreyer HC, Fry CS, Glynn EL, Rasmussen BB. Nutritional and contractile regulation of human skeletal muscle protein synthesis and mTORC1 signaling. J Appl Physiol (1985). 2009 Apr;106(4):1374-84. doi: 10.1152/japplphysiol.91397.2008. Epub 2009 Jan 15. PMID 19150856
- [Result] Dickinson JM, Rasmussen BB. Essential amino acid sensing, signaling, and transport in the regulation of human muscle protein metabolism. Curr Opin Clin Nutr Metab Care. 2011 Jan;14(1):83-8. doi: 10.1097/MCO.0b013e3283406f3e. PMID 21076294
- [Result] Fry CS, Rasmussen BB. Skeletal muscle protein balance and metabolism in the elderly. Curr Aging Sci. 2011 Dec;4(3):260-8. doi: 10.2174/1874609811104030260. PMID 21529326
- [Result] Walker DK, Dickinson JM, Timmerman KL, Drummond MJ, Reidy PT, Fry CS, Gundermann DM, Rasmussen BB. Exercise, amino acids, and aging in the control of human muscle protein synthesis. Med Sci Sports Exerc. 2011 Dec;43(12):2249-58. doi: 10.1249/MSS.0b013e318223b037. PMID 21606874
- [Result] Bell JA, Fujita S, Volpi E, Cadenas JG, Rasmussen BB. Short-term insulin and nutritional energy provision do not stimulate muscle protein synthesis if blood amino acid availability decreases. Am J Physiol Endocrinol Metab. 2005 Dec;289(6):E999-1006. doi: 10.1152/ajpendo.00170.2005. Epub 2005 Jul 19. PMID 16030064
- [Result] Bell JA, Volpi E, Fujita S, Cadenas JG, Sheffield-Moore M, Rasmussen BB. Skeletal muscle protein anabolic response to increased energy and insulin is preserved in poorly controlled type 2 diabetes. J Nutr. 2006 May;136(5):1249-55. doi: 10.1093/jn/136.5.1249. PMID 16614412
- [Result] Dreyer HC, Fujita S, Cadenas JG, Chinkes DL, Volpi E, Rasmussen BB. Resistance exercise increases AMPK activity and reduces 4E-BP1 phosphorylation and protein synthesis in human skeletal muscle. J Physiol. 2006 Oct 15;576(Pt 2):613-24. doi: 10.1113/jphysiol.2006.113175. Epub 2006 Jul 27. PMID 16873412
- [Result] Fujita S, Rasmussen BB, Bell JA, Cadenas JG, Volpi E. Basal muscle intracellular amino acid kinetics in women and men. Am J Physiol Endocrinol Metab. 2007 Jan;292(1):E77-83. doi: 10.1152/ajpendo.00173.2006. Epub 2006 Aug 8. PMID 16896165
- [Result] Fujita S, Rasmussen BB, Cadenas JG, Drummond MJ, Glynn EL, Sattler FR, Volpi E. Aerobic exercise overcomes the age-related insulin resistance of muscle protein metabolism by improving endothelial function and Akt/mammalian target of rapamycin signaling. Diabetes. 2007 Jun;56(6):1615-22. doi: 10.2337/db06-1566. Epub 2007 Mar 9. PMID 17351147
- [Result] Fujita S, Dreyer HC, Drummond MJ, Glynn EL, Cadenas JG, Yoshizawa F, Volpi E, Rasmussen BB. Nutrient signalling in the regulation of human muscle protein synthesis. J Physiol. 2007 Jul 15;582(Pt 2):813-23. doi: 10.1113/jphysiol.2007.134593. Epub 2007 May 3. PMID 17478528
- [Result] Fujita S, Abe T, Drummond MJ, Cadenas JG, Dreyer HC, Sato Y, Volpi E, Rasmussen BB. Blood flow restriction during low-intensity resistance exercise increases S6K1 phosphorylation and muscle protein synthesis. J Appl Physiol (1985). 2007 Sep;103(3):903-10. doi: 10.1152/japplphysiol.00195.2007. Epub 2007 Jun 14. PMID 17569770
- [Result] Dreyer HC, Glynn EL, Lujan HL, Fry CS, DiCarlo SE, Rasmussen BB. Chronic paraplegia-induced muscle atrophy downregulates the mTOR/S6K1 signaling pathway. J Appl Physiol (1985). 2008 Jan;104(1):27-33. doi: 10.1152/japplphysiol.00736.2007. Epub 2007 Sep 20. PMID 17885021
- [Result] Glynn EL, Lujan HL, Kramer VJ, Drummond MJ, DiCarlo SE, Rasmussen BB. A chronic increase in physical activity inhibits fed-state mTOR/S6K1 signaling and reduces IRS-1 serine phosphorylation in rat skeletal muscle. Appl Physiol Nutr Metab. 2008 Feb;33(1):93-101. doi: 10.1139/H07-149. PMID 18347658
- [Result] Dreyer HC, Drummond MJ, Pennings B, Fujita S, Glynn EL, Chinkes DL, Dhanani S, Volpi E, Rasmussen BB. Leucine-enriched essential amino acid and carbohydrate ingestion following resistance exercise enhances mTOR signaling and protein synthesis in human muscle. Am J Physiol Endocrinol Metab. 2008 Feb;294(2):E392-400. doi: 10.1152/ajpendo.00582.2007. Epub 2007 Dec 4. PMID 18056791
- [Result] Drummond MJ, Glynn EL, Lujan HL, Dicarlo SE, Rasmussen BB. Gene and protein expression associated with protein synthesis and breakdown in paraplegic skeletal muscle. Muscle Nerve. 2008 Apr;37(4):505-13. doi: 10.1002/mus.20976. PMID 18236467
- [Result] Drummond MJ, Fujita S, Abe T, Dreyer HC, Volpi E, Rasmussen BB. Human muscle gene expression following resistance exercise and blood flow restriction. Med Sci Sports Exerc. 2008 Apr;40(4):691-8. doi: 10.1249/MSS.0b013e318160ff84. PMID 18317375
- [Result] Drummond MJ, Bell JA, Fujita S, Dreyer HC, Glynn EL, Volpi E, Rasmussen BB. Amino acids are necessary for the insulin-induced activation of mTOR/S6K1 signaling and protein synthesis in healthy and insulin resistant human skeletal muscle. Clin Nutr. 2008 Jun;27(3):447-56. doi: 10.1016/j.clnu.2008.01.012. Epub 2008 Mar 14. PMID 18342407
- [Result] Drummond MJ, Dreyer HC, Pennings B, Fry CS, Dhanani S, Dillon EL, Sheffield-Moore M, Volpi E, Rasmussen BB. Skeletal muscle protein anabolic response to resistance exercise and essential amino acids is delayed with aging. J Appl Physiol (1985). 2008 May;104(5):1452-61. doi: 10.1152/japplphysiol.00021.2008. Epub 2008 Mar 6. PMID 18323467
- [Result] Dreyer HC, Drummond MJ, Glynn EL, Fujita S, Chinkes DL, Volpi E, Rasmussen BB. Resistance exercise increases human skeletal muscle AS160/TBC1D4 phosphorylation in association with enhanced leg glucose uptake during postexercise recovery. J Appl Physiol (1985). 2008 Dec;105(6):1967-74. doi: 10.1152/japplphysiol.90562.2008. Epub 2008 Oct 9. PMID 18845784
- [Result] Drummond MJ, Rasmussen BB. Leucine-enriched nutrients and the regulation of mammalian target of rapamycin signalling and human skeletal muscle protein synthesis. Curr Opin Clin Nutr Metab Care. 2008 May;11(3):222-6. doi: 10.1097/MCO.0b013e3282fa17fb. PMID 18403916
- [Derived] Borack MS, Dickinson JM, Fry CS, Reidy PT, Markofski MM, Deer RR, Jennings K, Volpi E, Rasmussen BB. Effect of the lysosomotropic agent chloroquine on mTORC1 activation and protein synthesis in human skeletal muscle. Nutr Metab (Lond). 2021 Jun 12;18(1):61. doi: 10.1186/s12986-021-00585-w. PMID 34118944
- [Derived] Graber TG, Borack MS, Reidy PT, Volpi E, Rasmussen BB. Essential amino acid ingestion alters expression of genes associated with amino acid sensing, transport, and mTORC1 regulation in human skeletal muscle. Nutr Metab (Lond). 2017 May 11;14:35. doi: 10.1186/s12986-017-0187-1. eCollection 2017. PMID 28503190
- [Derived] Dickinson JM, Gundermann DM, Walker DK, Reidy PT, Borack MS, Drummond MJ, Arora M, Volpi E, Rasmussen BB. Leucine-enriched amino acid ingestion after resistance exercise prolongs myofibrillar protein synthesis and amino acid transporter expression in older men. J Nutr. 2014 Nov;144(11):1694-702. doi: 10.3945/jn.114.198671. Epub 2014 Sep 3. PMID 25332468
- [Derived] Dickinson JM, Drummond MJ, Fry CS, Gundermann DM, Walker DK, Timmerman KL, Volpi E, Rasmussen BB. Rapamycin does not affect post-absorptive protein metabolism in human skeletal muscle. Metabolism. 2013 Jan;62(1):144-51. doi: 10.1016/j.metabol.2012.07.003. Epub 2012 Sep 6. PMID 22959478